CLINICAL TRIAL: NCT02720679
Title: Investigation of the Genetics of Hematologic Diseases
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Boston Children's Hospital (Other); University of Memphis (Other); Monroe Carell Jr. Children's Hospital at Vanderbilt (Other); Baylor College of Medicine (Other); Children's Hospital of Philadelphia (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: INSIGHT-HD
Record Dates: First submitted 2016-03-16; First posted 2016-03-28 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Bone Marrow Failure Syndromes; Erythrocyte Disorder; Leukocyte Disorder; Hemostasis; Blood Coagulation Disorder; Sickle Cell Disease; Dyskeratosis Congenita; Diamond-Blackfan Anemia; Congenital Thrombocytopenia; Severe Congenital Neutropenia; Fanconi Anemia; Myelodysplastic Syndromes; Myeloproliferative Diseases
Keywords: Genetics; Whole genome sequencing; Pediatrics and hematology
MeSH Terms: conditions — Bone Marrow Failure Disorders; Leukocyte Disorders; Blood Coagulation Disorders; Anemia, Sickle Cell; Dyskeratosis Congenita; Anemia, Diamond-Blackfan; Neutropenia, Severe Congenital, Autosomal Recessive 3; Fanconi Anemia; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples, bone marrow aspirate samples, nail clippings, urine, saliva, buccal smears and hair follicles, left over tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Participants will be (1) individuals with a non-malignant hematologic disorder confirmed or suspected to have a genetic basis, and (2) affected and unaffected family members of those individuals who are willing to provide clinical data and undergo genetic testing.

SUMMARY:
The purpose of this study is to collect and store samples and health information for current and future research to learn more about the causes and treatment of blood diseases. This is not a therapeutic or diagnostic protocol for clinical purposes. Blood, bone marrow, hair follicles, nail clippings, urine, saliva and buccal swabs, left over tissue, as well as health information will be used to study and learn about blood diseases by using genetic and/or genomic research. In general, genetic research studies specific genes of an individual; genomic research studies the complete genetic makeup of an individual.

It is not known why many people have blood diseases, because not all genes causing these diseases have been found. It is also not known why some people with the same disease are sicker than others, but this may be related to their genes. By studying the genomes in individuals with blood diseases and their family members, the investigators hope to learn more about how diseases develop and respond to treatment which may provide new and better ways to diagnose and treat blood diseases.

Primary Objective:

* Establish a repository of DNA and cryopreserved blood cells with linked clinical information from individuals with non-malignant blood diseases and biologically-related family members, in conjunction with the existing St. Jude biorepository, to conduct genomic and functional studies to facilitate secondary objectives.

Secondary Objectives:

* Utilize next generation genomic sequencing technologies to Identify novel genetic alternations that associate with disease status in individuals with unexplained non-malignant blood diseases.
* Use genomic approaches to identify modifier genes in individuals with defined monogenic non-malignant blood diseases.
* Use genomic approaches to identify genetic variants associated with treatment outcomes and toxicities for individuals with non-malignant blood disease.
* Use single cell genomics, transcriptomics, proteomics and metabolomics to investigate biomarkers for disease progression, sickle cell disease (SCD) pain events and the long-term cellular and molecular effects of hydroxyurea therapy.
* Using longitudinal assessment of clinical and genetic, study the long-term outcomes and evolving genetic changes in non-malignant blood diseases.

Exploratory Objectives

* Determine whether analysis of select patient-derived bone marrow hematopoietic progenitor/stem (HSPC) cells or induced pluripotent stem (iPS) cells can recapitulate genotype-phenotype relationships and provide insight into disease mechanisms.
* Determine whether analysis of circulating mature blood cells and their progenitors from selected patients with suspected or proven genetic hematological disorders can recapitulate genotype-phenotype relationships and provide insight into disease mechanisms.

DETAILED DESCRIPTION:
Participants will be individuals (proband) receiving therapy or expert consultation regarding a non-malignant hematologic disorder. We propose to use genomics, transcriptomics, proteomics and metabolomic analysis coupled with family linkage studies to identify causal mutations in individuals with undefined hematologic disorders and to characterize genetic modifiers of defined monogenic blood diseases.

A detailed medical history will be obtained, including demographic information for each proband. For each identified biologically related family member, a medical history questionnaire will be obtained. The family history and pedigree will be reviewed in conjunction with a geneticist/genetic counselor. The implications of genetic testing will be explained. If participants consent for future contact, this will take place annually for updates on medical and family history.

All probands will provide peripheral blood samples, and probands who are undergoing a bone marrow aspirate/biopsy for clinical purposes will provide additional aspirates. Biological family members will provide peripheral blood samples as a source for DNA.

ELIGIBILITY:
Inclusion Criteria:

* An individual (proband) receiving therapy or expert consultation regarding a non-malignant hematologic disorder, MDS or MPN.
* A biologically-related individual to the identified proband to include: first, second or third degree relatives.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be (1) individuals with a non-malignant hematologic disorder confirmed or suspected to have a genetic basis, and (2) affected and unaffected family members of those individuals who are willing to provide clinical data and undergo genetic testing.
Sampling Method: Non-Probability Sample
Enrollment: 1716 (Estimated)
Dates: Start 2016-06-17 (Actual); Primary Completion 2040-07 (Estimated); Study Completion 2050-07 (Estimated)

PRIMARY OUTCOMES:
Percent of participants who agree to participate | Day 1, at enrollment
  It is estimated that approximately 30% of participants (proband) approached for this study will agree to participate and that each proband will have approximately five biologically-related family members who agree to participate.

SECONDARY OUTCOMES:
Number by type of inherited genetic aberrations associated with hematologic disorders | Blood drawn at study entry, yearly and as needed until July 2050; and/or bone marrow aspirate at study entry, yearly and as needed until July 2050
  Germ-line DNA samples from study participants will be extracted and analyzed in order to identify inherited genetic aberrations associated with hematologic disorders. Specific modalities of genomic testing will be case specific. Relevant tests may involve SNP arrays to assess copy number variation, WGS, WES, targeted sequencing of specific candidate genes, DNA sequencing, RNA-sequencing, X-chromosome inactivation studies, ChIP sequencing and/or other tests. Genetic linkage analyses may be performed using a variety of technologies including high-density SNP arrays, WGS and specific analysis of selected target genes in validation studies.
Number by type of modifier genes | Blood drawn at study entry, yearly, and as needed until July 2050; and/or bone marrow aspirate at study entry, yearly and as needed until July 2050.
  Investigators seek to identify modifier genes in individuals in the study population. Methods of analysis will be similar to those for Outcome Measure #2.
Number by type of genetic variants | Blood drawn at study entry, yearly and as needed until July 2050; and/or bone marrow aspirate at study entry, yearly and as needed until July 2050.
  Investigators seek to identify genetic variants associated with treatment outcomes and toxicities in the study population. Methods of analysis will be similar to those for Outcome Measure #2.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Wlodarski, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: INSIGHT-HD Study Summary — http://www.stjude.org/treatment/clinical-trials/insight-hd-hematological-disorder.html
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols